CLINICAL TRIAL: NCT04957706
Title: Diagnostic Study of Anterior Cruciate Ligament Rupture With Anterior Drawer Test at 90° of Hip Flexion
Brief Title: Diagnostic Study of ACL Rupture With Anterior Drawer Test at 90° of Hip Flexion
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2019116
Record Dates: First submitted 2021-06-27; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-06

CONDITIONS: Anterior Cruciate Ligament Rupture
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute injury: injury ≤ 2 months
  Interventions: Diagnostic Test: anterior drawer test at 90° of hip flexion; Diagnostic Test: Lachman test; Diagnostic Test: anterior drawer test; Diagnostic Test: pivot-shift test
- Chronic injury: injury > 2 months
  Interventions: Diagnostic Test: anterior drawer test at 90° of hip flexion; Diagnostic Test: Lachman test; Diagnostic Test: anterior drawer test; Diagnostic Test: pivot-shift test

INTERVENTIONS:
Diagnostic Test: anterior drawer test at 90° of hip flexion — anterior drawer test at 90° of hip flexion
Diagnostic Test: Lachman test — Lachman test
Diagnostic Test: anterior drawer test — anterior drawer test
Diagnostic Test: pivot-shift test — pivot-shift test

SUMMARY:
For patients with anterior cruciate ligament rupture, the existing physical examinations have certain limitations. The researchers improved the traditional anterior drawer test in clinical work, maintained the flexion of the knee and flexion of the hip, and observed the displacement of the tibia. Good diagnostic effect, but no research statistics. The purpose of this study is to explore the effectiveness of the 90° of hip flextion anterior drawer test in the diagnosis of anterior cruciate ligament rupture.

DETAILED DESCRIPTION:
A total of 300 hospitalized patients who were diagnosed with anterior cruciate ligament rupture by MR and prepared for anterior cruciate ligament reconstruction were included, of which 150 cases were injured in the acute phase (within 2 months after the injury) and the chronic phase (more than 2 months after the injury). After the patient was admitted to the hospital, the patients were sequentially subjected to the 90° anterior drawer test, Lachman test, pivot-shift test, and anterior drawer test. The examination results were recorded. Compare the effectiveness of different physical examinations in diagnosing the anterior cruciate ligament. The patient's age, gender, injury time, BMI, the type of ACL rupture in the surgical records, and whether meniscus or cartilage damage were combined were counted. Regression analysis was used to evaluate the influencing factors of the modified anterior drawer test to correctly diagnose the rupture of the ACL.

ELIGIBILITY:
Inclusion Criteria:

* （1）ages between 18 and 60 years old. (2) Inpatients diagnosed with unique anterior cruciate ligament rupture and ready for anterior cruciate ligament reconstruction. (3) no combined injuries.

Exclusion Criteria:

* (1) The patient is younger than 18 years old or older than 60 years old, (2) multiple ligament injuries of the knee joint are suspected, and (3) combined fractures are suspected.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patient are from Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
anterior drawer test at 90° of hip flexion | 1 week after injury
  anterior drawer test at 90° of hip flexion

CONTACTS AND LOCATIONS:
Overall Officials: yingfang ao, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided